CLINICAL TRIAL: NCT05878379
Title: The Effects of a Dietary Iron Program on Iron Status and Cognitive Function Amoung School Children in Phatthalung Province, Southern Thailand
Brief Title: Effect of a Dietary Iron Program on Iron Status and IQ in Children in Phatthalung Province, Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUPH 2018-048
Record Dates: First submitted 2023-04-05; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Iron Deficiency, Anaemia in Children
Keywords: Iron deficiency; Iron status; Cognitive function; education
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: Quasi-experimental (pre-test post-test) design with follow-up / Behavioral intervention, based on the Health Belief Model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Iron Program (Experimental): The dietary iron program was administered from weeks 2 to 15 in between pre-test and post-test measurements
  Interventions: Behavioral: Dietary Iron Program

INTERVENTIONS:
Behavioral: Dietary Iron Program — Teachers Lesson 1: Discuss about causes, prevention and effects of anemia and ID, dietary iron, dietary enhancers and inhibitors of iron absorption, and school lunch menu Lesson 2: Participate in and observe how to teach children in an iron curriculum
  Caregivers Lesson 1: Presentation and group talk about causes, prevention, and effects of anemia and ID, dietary iron, and dietary enhancers and inhibitors of iron absorption Lesson 2: Discuss benefits and barriers of changing to an iron-rich meal at home Lesson 3: Cooking class for preparing an iron-rich meal at home (2 times) Lesson 4: Home visit
  Children Lesson 1: Group talk about causes and effects of anemia and ID Games: "Where are you from?" Lesson 2: Presentation and group talk about dietary iron, and dietary enhancers and inhibitors of iron absorption, and iron-rich food Games: "What is the winner?" Assignment: Market assignment Lesson 3: Cooking class (2 times)

SUMMARY:
Iron deficiency (ID) continues to be one of the most prevalent disorders, which can adversely affect cognitive ability in childhood. Our aim was to determine the effect of a dietary iron education program (DIP) on children's iron status and intelligence quotient (IQ) score. This pre-test (week 1) post-test (week 16) quasi-experimental study with follow-up (week 18) utilized constructs from the Health Belief Model. Children and caregivers participated in the DIP which incorporated group talks, presentations, brainstorming, game-based learning and cooking sessions from weeks 2-15. Knowledge of ID and dietary iron, perceived susceptibility and severity, benefits and barriers for changing behavior, dietary intake, iron status and IQ score were determined at all timepoints (weeks 1, 16, and 18).

DETAILED DESCRIPTION:
1. Objective The objective of this study was to determine whether an education-based dietary iron program that involved school teachers, parents and children could increase iron status and intelligence quotient (IQ) score in a group of schoolchildren.
2. Methods

2.1 Study design A quasi-experimental study (pre-test post-test design with follow-up) was used in this study that was based on the Health Belief Model as its theoretical framework.

2.2 Study Setting and Participants Child-parent/caregiver dyads were recruited from one purposively selected government-administered primary school in Phatthalung province. Schools were not involved in any other programs, located in a rural area, and had at least 200 children studying in grades 4-5. Hookworm screening was done 6 weeks before program implementation by the local government screening program. All children who were studying in grades 4-5 in the selected school were invited to participate. Out of 190 children, 34 children who were mildly anemic were enrolled in the study, together with their parents/caregivers. Sample size was calculated based on serum ferritin concentrations among school-aged children from a study by Rahman et al. [17]. Informed written consent was obtained from child-parent/caregiver dyads prior to program implementation.

2.3 Procedure for the intervention The Health Belief Model underpinned the development of the dietary iron program, which focused on the importance of adequate dietary iron consumption and emphasized prevention of iron deficiency (ID) and iron deficiency anemia (IDA). It was implemented from weeks 2 to 15 of the study. Child-parent/caregiver dyads and teachers received an ID/IDA booklet that included information about anemia, causes of ID, iron-rich food, iron concentration in traditional foods, dietary enhancers and inhibitors of iron absorption, and recipes for iron-rich local and culturally appropriate meals for teachers, parents/caregivers and children, as part of the dietary iron program.

Teachers who were involved in school lunch design participated for discussing and planning iron-rich school lunch menus, and observed teaching and learning process with the use of media and games during the iron lessons for children. Four lessons were conducted for parents/caregivers. The first lesson was discussion that addressed parental perceptions about children's susceptibility to ID and IDA and the severity of ID and IDA concerning cognitive function. In the second lesson, parents/caregivers were asked to list the benefits and barriers for changing behavior with regards to preparing more iron-rich foods in the home. Then, the principal researcher invited parents/caregivers to brainstorm and share ways to overcome these barriers. Cooking classes for preparing iron-rich meals at home were conducted. Parents/caregivers voted for two iron-rich meals that they wanted to cook and then they prepared and cooked them in the classes. For the final lesson, the principal researcher visited each parent/caregiver to discuss the barriers they faced when trying to incorporate more iron-rich meals into their child's diet at home. Three lessons were conducted for the children, one per month. In the first lesson, group talks and games were used to engage the children about the causes and effects of ID and IDA. The second lesson focused on iron-rich food. After that, the children partook in games that entailed writing names of food ingredients that contained iron and circling pictures of iron-rich foods, and describing the sensations associated with consuming these foods. Both positive and negative answers from children were selected for discussion, and approaches for consuming more iron-rich food were brainstormed. A market assignment was set to help the children remember the names of iron-rich food and recognize the foods when they visited a market with their parents. The last lesson was a cooking class. After each cooking class finished, the researcher and a teacher encouraged them to eat this meal together.

2.4 Measurement outcomes The main outcome for this study was the effect of an education-based dietary iron program on iron status and intelligence quotient (IQ) score among children before program implementation (week 1) and at week 16 (immediately after program implementation) and at 18 weeks (follow-up appointment to determine the sustainability of the intervention). All of the outcome variables were measured at different time points. Children's knowledge towards ID and IDA was determined using a questionnaire, while children's iron intake was estimated by using three days of 24-hour recalls (2 school days and 1 weekend day). Portion sizes were estimated by using household portion sizes (rice-serving spoon, tablespoon, teaspoon and glass). IQ score was measured by a trained child psychologist by using the Standard Progressive Matrices (SPM) parallel version. Iron status was determined from blood samples drawn by medical technologists in the first-aid rooms. Concentration of hemoglobin, serum ferritin and serum C-reactive protein were measured by laboratory staff at hematology laboratory at N-health laboratory, Bangkok Dusit Medical Service Hospital (BDMS), Songkla province, using the hemoglobin assay kit (Colorimetric), chemiluminescent immunoassay (CMIA) and high-sensitivity C-reactive protein methods, respectively. Iron status was defined iron-replete: hemoglobin >115 g/l and serum ferritin level > 30 µg/l; anemia: hemoglobin <115 g/l and serum ferritin level >30 µg/l; mild-moderate iron depletion with anemia: hemoglobin 80-114 g/l and serum ferritin level <30 µg/l.; mild iron depletion without anemia: serum ferritin level < 30 µg/l and hemoglobin>115 g/l. In addition, parents/caregivers were assessed by using a questionnaire toward knowledge and perceptions consisted of perceived susceptibility, severity, benefits and barriers in relation to ID and IDA.

2.5 Data Analysis Data from questionnaires were recorded using EpiData version 3.1, while 24-hour dietary recall data were entered into INMUCAL V3, which is a nutrient composition database of dietary items commonly consumed in Thailand. Portion sizes were converted into grams before entering data, and energy and nutrient intakes were calculated. Statistical analysis was carried out by using SPSS version 18. Frequencies, percentage, mean (SD) and median (25th-75th percentile) were calculated for demographic characteristics of participant knowledge, perceptions, iron intake, iron status, and IQ score. The One-Way Repeated Measures ANOVA and Friedman's Two-Way Analysis of Variance by Ranks were used to compare mean differences in knowledge score and perception score of IDA and ID prevention among parents/caregivers, total iron intake, heme iron intake, non-heme iron intake, iron status and IQ score among children at different time points. The Monte Carlo exact test was used to compare the number of children in grades 4-5 who met/did not meet the Thai DRI for iron at pre-test, post-test and follow-up. Differences were considered to be significantly different when p<0.05.

2.6 Ethical approval The study was granted ethical approval by the Committee of the Ethical Review for Human Research, Faculty of Public Health, Mahidol University Thailand 9 March 2018 (COA. No. MUPH 2018-048).

ELIGIBILITY:
Inclusion Criteria:

* Children who were studying in grades 4 and 5 of the selected school

Exclusion Criteria:

* Severe illness, including severe anemia (hemoglobin <4.96 mmol/L or <80 g/L)
* Post-menarche
* Use of vitamin or mineral supplements up to 30 days before program implementation

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Iron Status | Change from baseline (week 1) to post-test (week 16), and change from post-test (week 16) to follow-up (week 18)
  For outcome 1, individuals were categorized as either: (1.) iron replete, (2.) Iron deficient, (3.) Iron deficient with mild-moderate anemia (4.) mild-moderately anemic

SECONDARY OUTCOMES:
Intelligence quotient (IQ) score | Change from baseline (week 1) to post-test (week 16), and change from post-test (week 16) to follow-up (week 18)
  Outcome 2 was measured as the number of IQ points (continuous data)

CONTACTS AND LOCATIONS:
Overall Officials: Witchada Simla, MSc, Principal Investigator — Thaksin University (Phatthalung Campus), Thailand
Locations (1):
- Ms Witchada Simla, Phatthalung, Phattalung Province, Thailand

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared with researchers outside of the research team.